CLINICAL TRIAL: NCT06323109
Title: Ultrasound Imaging for the Assessment of Lower Urinary Tract Symptoms
Brief Title: US Imaging for the Assessment of LUTS
Status: Recruiting | Type: Observational
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: Wisconsin Partnership Program (Other)
Responsible Party: Sponsor
Other Study IDs: 2023-1331; A196200 (Other: UW Madison); Protocol Version 12/19/24 (Other: UW Madison)
Record Dates: First submitted 2024-03-14; First posted 2024-03-21 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Lower Urinary Tract Symptoms; BPH
MeSH Terms: conditions — Lower Urinary Tract Symptoms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (2):
- Healthy Controls: Age-matched healthy men with no lower urinary tract symptoms
  Interventions: Device: MRI-UDS; US-UDS; MCUD
- Known BPH/LUTS: Adult men diagnosed with BPH/LUTS
  Interventions: Device: MRI-UDS; US-UDS; MCUD

INTERVENTIONS:
Device: MRI-UDS; US-UDS; MCUD — Imaging procedures will include a comprehensive protocol of dynamic MRI, 3D ultrasound and MCUD to evaluate and validate this entirely novel methodology.

SUMMARY:
The purpose of this research is to develop an ultrasound (US) based urodynamics (UDS) evaluation of voiding based on successful magnetic resonance imaging (MRI)-UDS evaluation. Both US and MRI are non-invasive imaging techniques, but US is a more cost-effective and widely available technology. 80 participants will be enrolled and will be on study for up to 2.5 hours (1.5 hour MRI and 1 hour US).

DETAILED DESCRIPTION:
The MRI - UDS technique provides voiding flow rates and bladder pressures which can be used to calculate the widely used metrics of obstruction (bladder outlet obstruction index, BOOI) and contractility (bladder contractility index, BCI). In a preliminary study, values for maximum flow (Qmax) and detrusor pressure at maximum flow (PdetQmax) were obtained from MRI-UDS for patients with BPH/LUTS. These results closely correlated with multichannel urodynamics (MCUD).

Men with BPH/LUTS and age-matched controls will undergo a comprehensive protocol of dynamic MRI, 3D ultrasound and multi-channel urodynamics (MCUD) to evaluate and validate this novel methodology.

Specific aims include:

Aim 1. Develop an ultrasound/CFD based urodynamics (US-UDS) method. A protocol combining 3D US imaging and CFD analysis will be developed. This approach will be validated both in vitro and in vivo, first in an anatomically realistic model and then in control human subjects.

Aim 2. Establish the accuracy of voiding metrics determined with ultrasound urodynamics (US-UDS). MCUD, MRI-UDS and the new US-UDS protocols will all be performed to evaluate voiding in patients with BPH/LUTS and healthy controls. Urodynamic metrics derived from ultrasound will be compared to those obtained from the reference clinical standard MCUD and MRI-UDS.

Aim 3. Develop an optical velocimetry methods that allows the non-invasive quantification of urine velocity while voiding. A setup of high speed cameras will be assembled and utilized to optically image the voiding stream in all subjects recruited for aims 1 and 2.

ELIGIBILITY:
Inclusion Criteria: Patients with BPH/LUTS

* Age 18-80 years old
* Diagnosed with BPH/LUTS with or without obstruction

Exclusion Criteria:

* Patients with contraindication to MRI and/or GBCA contrast agent. Diabetic subjects will not receive contrast.
* History of overt neurologic disease other than diabetic neuropathy, urinary tract infection within the last 4 weeks or recent history of urinary retention (within the last 4 weeks).

Inclusion Criteria: Healthy Volunteers

- Age 18-80 years old not experiencing any symptoms consistent with LUTS

Exclusion Criteria:

* Patients with contraindication to MRI and/or GBCA contrast agent.
* Currently taking medications with known effects on the bladder, overt neurologic disease other than diabetic neuropathy, urinary tract infection within the last 4 weeks or urinary retention symptoms.

Ages: 18 Years to 80 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Patients targeted for enrollment will be based on the diagnosis of BPH.
Study Population: 1. Men diagnosed with BPH/LUTS
  2. Healthy volunteers
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2023-11-28 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
MRI Urodynamics - Change in Bladder Volume | Research visit 1 day
  MRI-based CFD technique (MRI - UDS) provides voiding flow rates and bladder pressures which can be used to calculate the widely used metrics of obstruction (bladder outlet obstruction index, BOOI) and contractility (bladder contractility index, BCI).
  Bladder volumes are quantified from the time resolved volumetric data acquired during the void event in each patient.
  The outcomes from the MRI based CFD simulations of the voiding event are urine velocity and pressure in the bladder and urethra at the different time points during the void.
MRI Urodynamics - Change in Urine Velocity | Research visit 1 day
  MRI-based CFD technique (MRI - UDS) provides voiding flow rates and bladder pressures which can be used to calculate the widely used metrics of obstruction (bladder outlet obstruction index, BOOI) and contractility (bladder contractility index, BCI). Flow rates are derived from the volume change of the bladder. Volumes are quantified from the time resolved volumetric data acquired during the void in each patient. Calculated flow rate is used to computationally estimate the pressure required to drive that flow using computational fluid dynamics.
  In summary, the outcome from the MRI acquisition is bladder volume as well as urethral anatomy during the void event. The outcomes from the MRI based CFD simulations of the voiding event are urine velocity and pressure in the bladder and urethra at the different time points during the void.
MRI Urodynamics - Change in Pressure | Research visit 1 day
  MRI-based CFD technique (MRI - UDS) provides voiding flow rates and bladder pressures which can be used to calculate the widely used metrics of obstruction (bladder outlet obstruction index, BOOI) and contractility (bladder contractility index, BCI). Flow rates are derived from the volume change of the bladder. Volumes are quantified from the time resolved volumetric data acquired during the void in each patient. Calculated flow rate is used to computationally estimate the pressure required to drive that flow using computational fluid dynamics.
  In summary, the outcome from the MRI acquisition is bladder volume as well as urethral anatomy during the void event. The outcomes from the MRI based CFD simulations of the voiding event are urine velocity and pressure in the bladder and urethra at the different time points during the void.
Bladder outlet obstruction index (BOOI) | Research visit 1 day
  Bladder outlet obstruction index (BOOI): A metric of obstruction calculated from MRI flow rates and bladder pressures then compared to US values.
  BOOI, is derived from the equation PdetQmax - 2Qmax. Scores: <20 means unobstructed, 20-40 means equivocol, >40 means obstructed.
Bladder contractility index (BOI) | Research visit 1 day
  Bladder contractility index (BOI): a metric of bladder contractility calculated from MRI flow rates and bladder pressures then compared to US values.
  BOI is derived from the equation PdetQmax + 5Qmax. Scores: <100 means weak, 100-150 menas normal, >150 means strong.
International Prostate Symptom Score (IPSS) | Research visit 1 day
  The IPSS is a validated global questionnaire used to assess the degree of "bother" from benign prostatic hyperplasia symptoms based on the answers to 7 questions concerning urinary symptoms. Each question is assigned points from 0 to 5 indicating increasing severity of the particular symptom. The voiding score is the sum of the responses to 4 questions relating to urination (incomplete emptying, intermittency, weak stream and straining) and ranges from 0 to 20 (asymptomatic to very symptomatic).

CONTACTS AND LOCATIONS:
Overall Officials: Alejandro Roldan-Alzate, PhD, Principal Investigator — UW Department of Mechanical Engineering and Radiology
Locations (1):
- University of Wisconsin, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No